CLINICAL TRIAL: NCT03598309
Title: Phase II Trial of Investigational Agents to Modulate Intermediate Endpoint Biomarkers, Including Pulmonary Nodules, in Former and Current Smokers
Brief Title: Phase II Trial to Modulate Intermediate Endpoint Biomarkers in Former and Current Smokers
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: James and Esther King Biomedical Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MCC-19622; 8JK03 (Other: James & Esther King Biomedical Research Group)
Record Dates: First submitted 2018-07-13; First posted 2018-07-26 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Lung Diseases; Lung Cancer, Protection Against
Keywords: Lung RADS 3; Lung nodule; Lung cancer risk; Chemoprevention
MeSH Terms: conditions — Lung Diseases; Lung Neoplasms | interventions — Diarylheptanoids; Omacor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Curcumin C3 complex® +Lovaza® (Active Comparator): Group A:
  4 grams Lovaza®, 2 grams twice a day (BID). 2 grams by mouth daily, AM and PM 8,000 mgs CUR Curcumin C3 complex® tablets, divided into 2 doses. 4 grams by mouth, twice a day, AM and PM.
  Interventions: Drug: Curcumin C3 complex®; Drug: Lovaza®
- Curcumin C3 complex® +Lovaza® +Placebo (Active Comparator): Group B:
  2 grams Lovaza®, 1 gram twice a day, AM and PM. 4,000 mgs CUR Curcumin C3 complex® tablets, 2,000 mgs twice a day, AM and PM.
  1 placebo capsule twice a day, AM and PM.
  Interventions: Drug: Curcumin C3 complex®; Drug: Lovaza®; Other: Placebo
- Placebo only (Active Comparator): Placebo: Two matching placebo capsules twice a day (BID), taken by mouth, AM and PM
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Curcumin C3 complex® — Groups A and B as outlined in study arm. Drug will be dispensed by investigational pharmacists and self-administered by the participants.
  Other Names: Curcuminoid
  Arms: Curcumin C3 complex® +Lovaza®; Curcumin C3 complex® +Lovaza® +Placebo
Drug: Lovaza® — Groups A and B as outlined in study arm. Drug will be dispensed by investigational pharmacists and self-administered by the participants.
  Other Names: Omega-3-Acid Ethyl Esters
  Arms: Curcumin C3 complex® +Lovaza®; Curcumin C3 complex® +Lovaza® +Placebo
Other: Placebo — Groups B and Placebo as outlined in study arm. Drug will be dispensed by investigational pharmacists and self-administered by the participants.
  Other Names: Pill with no drug or other active ingredients in it.
  Arms: Curcumin C3 complex® +Lovaza® +Placebo; Placebo only

SUMMARY:
The purpose of this study is to find out if an investigational combination drug called Lovaza (made with fish oils)+Curcumin C3 Complex (made from a root called curcumin) can help reduce the size of lung nodules. Researchers also want to find out if the combination of Lovaza+Curcumin C3 Complex is safe and tolerable.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 55 years of age or older
* Former smokers and current enrolled in LDCT lung cancer screening or those who are detected using a regular CT, and have Lung-RADS 3 category lesion(s), that would get a 6 month f/u LDCT or regular CT based on Lung-RADS recommendations or former and current smokers enrolled in LDCT lung cancer screening, or regular CT and have Lung-RADS 2 category lesions with part-solid or non-solid lung nodule ≥4mm mean diameter detected during screening LDCT or regular CT scans
* History of cigarette smoking with ≥ 20 pack years
* All current smokers should accept to receive smoking cessation
* Eastern Cooperative Oncology Group (ECOG) Performance Status of less than or equal to 1
* Able to swallow study pills
* Able to undergo CT
* Not allergic to components of study agents
* Willing to discontinue current vitamin/mineral supplement use containing components of study agents. A standard multivitamin supplement provided for the study
* Willing to comply with proposed visit and treatment schedule
* Able to understand and willing to sign a written informed consent document
* Participants must have normal organ and marrow function
* Willing to use contraception during the intervention period of 6 months (males and females)
* Not pregnant or lactating nor planning to become pregnant or lactate during the 6 month study intervention period..

Exclusion Criteria:

* Invasive cancer diagnosis (excluding basal cell carcinoma or skin squamous cell carcinoma) diagnosed within the last 2 years
* Inability to undergo CT
* Newly diagnosed nodule meeting Lung-RADS 4 criteria
* Have taken doxycycline or tetracycline less than or equal to 2 weeks
* Females- pregnant or lactating (throughout the duration of intervention of 6 months)
* Unwilling to use effective form of birth control (Males and females) (throughout the duration of intervention of 6 months).

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Bronchial Nodule Size | 6 months post treatment
  Difference in the average change in bronchial nodule size from baseline to end of therapy at 6 months for each study arm. A lower size is taken to be the desired value for participants receiving study drug, assuming an increase in size for the placebo arm.
Rate of Nodules ≥4 mm | 6 months post treatment
  Number of nodules ≥4 mm per study arm, post treatment.

SECONDARY OUTCOMES:
Rate of Adherence | 6 months post treatment
  Rate of participant adherence per study arm. Proof of adherence based on study team pill counts, participant diet logs and pill logs at end of study, vs. data collected at midpoint.
Rate of Treatment Related Adverse Events (AEs) | Up to 30 days post treatment, approximately 7 months
  Safety of the combined agents (Curcumin C3 complex® + Lovaza®) at 2 dose arms vs. placebo as indicated by incidence of related adverse events and toxicities, monitored using Common Toxicity Criteria version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Nagi Kumar, Ph.D, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://www.moffitt.org/clinical-trials-research/clinical-trials/?gclid=EAIaIQobChMImIymzIa-9gIVAZ2GCh3uzAWJEAAYASAAEgI0ovD_BwE